CLINICAL TRIAL: NCT01743547
Title: THE EFFECTS OF YOGA ON QUALITY OF LIFE AMONG A POPULATION OF OVARIAN/ FALLOPIAN TUBE/ PRIMARY PERITONEAL CANCER PATIENTS RECEIVING CHEMOTHERAPY: A FEASIBILITY STUDY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigators concluded that it is not feasible due to the lack of participation and difficulty in recruiting patients.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Nikki Neubauer, Assistant Professor in Obstetrics and Gynecology, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NU12G05
Record Dates: First submitted 2012-11-30; First posted 2012-12-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Ovarian Cancer
Keywords: Women; Yoga; Ovarian Cancer; Lifestyle
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Yoga

ARMS (2):
- No Intervention; Arm A; Control Group (No Intervention): 24 subjects who declined yoga but agreed to data collection
- Active Comparator; Arm B; Intervention Group (Active Comparator): 24 subjects participating in 8 weeks of Yoga and agreed to data collection
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — Patients will be randomized to Yoga or control group. Those in Yoga intervention will receive 8 weekly yoga sessions.
  Arms: Active Comparator; Arm B; Intervention Group

SUMMARY:
This is a pilot study to establish the feasibility of an eight-week yoga intervention and to estimate the effect size on QoL in female patients with ovarian, fallopian tube and primary peritoneal malignancies receiving chemotherapy for the treatment of primary or recurrent cancer.

DETAILED DESCRIPTION:
The primary objective of this study was to determine the feasibility of implementing a yoga program among gynecologic cancer patients receiving chemotherapy. The investigators concluded that it is not feasible due to the lack of participation and difficulty in recruiting patients. Of 25 consented patients, 16 agreed to participate in the control arm, 9 agreed to participate in the Yoga classes. Three (3) of those 9 changed their minds and withdrew consent. Of the 6 remaining patients, only 3 attended at least 1 of the 8 classes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of epithelial ovarian/fallopian tube/primary peritoneal cancer
* Participant must be age 18 or older
* Participants must be 6 weeks post-surgery
* Participant must be currently receiving chemotherapy or beginning a regimen within the next four weeks
* Participant must be willing to attend the intervention sessions
* All subjects must have given signed, informed consent prior to registration in the study.

Exclusion Criteria:

* Participant has practiced yoga more than 4 times in the last year
* Participant has a surgical procedure scheduled during the 8 weeks that they would be part of the intervention
* Participant has an ECOG performance status less than or equal to two

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
All patients included in the study will be assessed for response to treatment; the primary outcome is change in QoL domains after yoga class intervention. Planned subgroup analysis: stratification by participation category | Total study duration is anticipated to require approximately 24 weeks
  Pilot study to establish the feasibility of a yoga program & estimate the effect size of a yoga intervention on QoL in patients with epithelial ovarian, fallopian tube & primary peritoneal cancer receiving chemotherapy for the treatment.The goal for each individual question on the questionnaire is to have a 90-95% completion rate. The validated instruments: FACT-O, FACIT-F, FACIT-Sp, CES-D, PROMIS, and PSQI will be scored according to their respective guidelines, and then paired t-tests will be used to compare the pre-yoga and post-yoga means.
  Participant completion will be recorded in one of three ways: complete, meaning the participant attended 5 or more yoga sessions and filled out all the required surveys; partially complete, meaning the participant attended 1-4 sessions, and/or did not fill out all the required surveys; and did not participate, meaning the participant attended 0 sessions. All analyses will be stratified for participation category.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States